CLINICAL TRIAL: NCT03342768
Title: A Smartphone Messaging Programme for Tobacco Industry Denormalisation - a Randomised Controlled Trial
Brief Title: An RCT of a Smartphone-based TID Programme
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Daniel Sai-Yin Ho, Principle investigator and associate professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: coshdrama
Record Dates: First submitted 2017-11-08; First posted 2017-11-17 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Tobacco Industry Denormalisation Beliefs; Tobacco-related Communications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TID (Experimental): Messages will be sent 1-2 times per week containing information that aims to denormalise the tobacco industry.
  Interventions: Other: Smartphone-based messages
- Sugar sweetened beverages (Other): Messages will be sent 1-2 times per week containing information on the adverse health effects of sugar sweetened beverages.
  Interventions: Other: Smartphone-based messages

INTERVENTIONS:
Other: Smartphone-based messages — For the TID arm, the messages' contents include the tobacco industry's (TI's) anti-smoking campaigns that made smoking more grown-up and more appealing to youth; the TI's role in smoking in movies; etc.
  For the sugar sweetened beverage (SSB) arm, the messages' contents include the disease conditions linked to SSBs, and the interference of sugar industry in scientific research.

SUMMARY:
The study aims to test the effect a smartphone-based intervention on primary school students and their parents' attitudes towards tobacco industry and their tobacco-related communications.

ELIGIBILITY:
Inclusion Criteria:

* Parents and children should all understand Chinese.
* Parents should have a smartphone and use WhatsApp (a smartphone-based app)

Exclusion Criteria:

* n/a

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2018-06-29 (Actual)

PRIMARY OUTCOMES:
TID beliefs in parents | 1 month
  Parents will report their opinions towards 4 sentences: 1) Tobacco companies are a respectable industry; 2) the tobacco industry does everything it can to get young people to smoke; 2) the tobacco industry use many tactics to resist tobacco control regulations; 4) the tobacco industry deceived the public for financial interests. All the 4 questions have 5 options from definitely yes to definitely no. The options will be recoded into 0-4 or 4-0, as appropriate, with higher scores indicating more negative attitudes towards the industry. A sum of scores from the 4 questions will be deemed a measurement of TID beliefs.
TID beliefs in children | 1 month
  Students will report their opinions towards 4 sentences: 1) Tobacco companies are a respectable industry; 2) the tobacco industry does everything it can to get young people to smoke; 2) the tobacco industry use many tactics to resist tobacco control regulations; 4) the tobacco industry deceived the public for financial interests. All the 4 questions have 5 options from definitely yes to definitely no. The options will be recoded into 0-4 or 4-0, as appropriate, with higher scores indicating more negative attitudes towards the industry. A sum of scores from the 4 questions will be deemed a measurement of TID beliefs.

SECONDARY OUTCOMES:
Tobacco related communication reported by parents | 1 month
  Parents will report whether they said the following to children in the past 30 days: 1) harm of smoking 2) harm of secondhand smoking 3) criticise smoking behaviour 4) approve tobacco control measures. Each of the messages will be analyse as a binary outcome.
Sugar sweetened beverage (SSB) related communication reported by parents | 1 month
  Parents will report whether they said the following to children in the past 30 days: 1) harm of SSB 2) certain kind of drinks contain sugar 3) don't drink or drink less SSB. Each of the messages will be analyse as a binary outcome.
Tobacco related communication reported by children | 1 month
  Students will report whether they heard the following from parents in the past 30 days: 1) harm of smoking 2) harm of secondhand smoking 3) criticize smoking behaviour 4) approve tobacco control measures. Each of the messages will be analyse as a binary outcome.
SSB related communication reported by children | 1 month
  Students will report whether they heard the following from parents in the past 30 days: 1) harm of SSB 2) certain kind of drinks contain sugar 3) don't drink or drink less SSB. Each of the messages will be analyse as a binary outcome.
Intention to smoke in children | 1 month
  Two questions will be used to assess this outcome: 1) do you think you will smoke in the next 12 months? 2) If one of your good friends offers you a cigarette, will you smoke it? Response options are definitely not/probably not/probably yes/definitely yes. Those choosing options other than "definitely not" for either of the questions will be deemed having intention to smoke; the other students will be deemed having no intention to smoke.
Home exposure to secondhand smoke in children reported by children | 1 month
  One question will be asked: 1) On how many of the past 7 days did someone smoke near you at home? (Options 0 day/1/2/3/4/5/6/7). The responses will dichotomised into a binary indicator of secondhand smoke exposure (no/any) and analysed as an outcome.
Home exposure to secondhand smoke in children reported by parents | 1 month
  One question will be asked: 1) On how many of the past 7 days did someone smoke near your children at home? (Options 0 day/1/2/3/4/5/6/7). The responses will dichotomised into a binary indicator of secondhand smoke exposure (no/any) and analysed as an outcome.
Parents' support for tobacco control | 1 month
  Parents will report their opinions towards 4 sentences: 1) government should adopt plain packaging; 2) government should impose stronger regulation on tobacco; 3) government should strengthen the prevention of the harm of tobacco. The options were strongly support/support/neutral/oppose/strongly oppose. The options will be recoded into 4-0, with higher scores indicating stronger support for tobacco control. A sum of scores from the 4 questions will be deemed a measurement of parents' support for tobacco control.
Negative attitude towards smoking in parents | 1 month
  Parents will be asked "your attitude towards smoking is" with options of very positive/positive/neutral/negative/very negative. The options will be dichotomised as very negative vs others (negative/neutral/positive/very positive) for analysis.
Negative attitude towards smoking in children | 1 month
  Children will be asked "your attitude towards smoking is" with options of very positive/positive/neutral/negative/very negative. The options will be dichotomised as very negative vs others (negative/neutral/positive/very positive) for analysis.
Past 7-day consumption of SSB and water in children reported by children | 1 month
  Children will be asked "On how many of the past 7 days did you drink SSBs?" and "On how many of the past 7 days did you drink water?" For both questions, the options were 0/1/2/3/4/5/6/7 days. These two variables will be analysed as both binary (No (0 day) vs any (1/2/3/4/5/6/7 days)) and continuous variables.
Past 7-day consumption of SSB and water in children reported by parents | 1 month
  Parents will be asked "On how many of the past 7 days did you drink SSBs?" and "On how many of the past 7 days did you drink water?" For both questions, the options were 0/1/2/3/4/5/6/7 days. These two variables will be analysed as both binary (No (0 day) vs any (1/2/3/4/5/6/7 days)) and continuous variables.

CONTACTS AND LOCATIONS:
Overall Officials: Sai Yin Ho, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Local primary schools, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided